CLINICAL TRIAL: NCT06188780
Title: Characteristics of (Unwanted) Use of Alcohol and Illicit Substances Among Patients Reporting After Sexual Violence in Ghent: a Mono-centric Prospective Observational Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2023-0076
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Drug-facilitated Sexual Assault
MeSH Terms: interventions — Urination; Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and/or urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- victims of DFSA: Every patients presenting at the sexual assault care centre with a suspicion of drug-assisted sexual assault
  Interventions: Diagnostic Test: urine/blood analysis with IA and LC-GCMS analysis

INTERVENTIONS:
Diagnostic Test: urine/blood analysis with IA and LC-GCMS analysis — urine/blood analysis with IA and LC-GCMS analysis
  Other Names: toxicology testing

SUMMARY:
This study aims at defining the patient characteristics and toxicological aspects of patients presenting at the sexual assault care centre with drugs-facilitated sexual assault.

DETAILED DESCRIPTION:
This study aims to map (un)voluntary use of alcohol and drugs among victims of sexual violence who present to the Care Centre after Sexual Violence at UZ Gent, referred to in English as Drug-Facilitated Sexual Assault (DFSA).

Sometimes substances are deliberately used to render a victim submissive (proactive DFSA), but it is also possible that people use substances themselves recreationally and later become victims of sexual violence (opportunistic DFSA).

Recent media reports of drinks in which psychogenic substances are involuntarily administered have become more frequent, after which people sometimes become victims of sexual violence. The public attention for this problem increased significantly recently. However, no clear data are currently available in Belgium on this problem.

Using a prospective observational study, we aim to map the incidence of (unwanted) use of alcohol and illegal substances among victims who report to the Care Centre after Sexual Violence in Ghent. The data - after obtaining informed consent - will be collected by means of (nurse-led) questionnaires and toxicological analyses on blood and urine samples. We envisage a two-year period for inclusion of patients, starting from 01/03/2023, running until 31/03/2025.

With these results, we want to estimate the proportion of sexual assault incidents in which the victim was incapacitated by voluntary or involuntary/unwanted use of alcohol or illicit substances (e.g. cannabis, GHB, cocaine, ...). To this end, we need to record data from all patients who present in order to estimate the denominator.

Every patients presenting at the sexual assault care centre with a suspicion of drug-assisted sexual assault, will be requested to take part in the study.

Patient data will be derived from the patient record, with regards to voluntary and unvoluntary administration of alcohol/illicit drugs/medication, previous medical history and symptoms.

Biological samples (blood and urine if <48h after event, and urine if between 48h and 96h after event) will be collected and analysed according to UNODC guidelines (Guidelines for the Forensic analysis of drugs facilitating sexual assault and other criminal acts) with IA and LC-GCMS testing.

ELIGIBILITY:
Inclusion Criteria:

* All patients (16+) who registered at the Care Center after Sexual Violence (=ZSG) in Ghent from 01/04/2023 until. 31/03/2025 and who were victims of sexual violence are eligible for inclusion in this study.

Exclusion Criteria:

* Reporting longer than 5 days after the sexual assault.
* Unable to undergo a forensic examination under the supervision of a forensic nurse due to, for example, collapse of consciousness or failure to give consent to do so.
* Not declaring proficiency in the language in which informed consent is offered (Dutch/English)
* Not agreeing to the informed consent.
* Not agreeing to collection and/or analysis of blood and urine.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Victims of DFSA (16+)
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
patient characteristics in objectivated DFSA | 19 months
  Characteristics of patients (medical history, symptoms) after DFSA
toxicology results in patients with DFSA | 19 months
  Results of toxicologic analysis in patients with DFSA

CONTACTS AND LOCATIONS:
Locations (1):
- ZSG UZ Gent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided